CLINICAL TRIAL: NCT03559036
Title: Impact of Activity-Dependent Plasticity on Bladder Function After Pediatric Spinal Cord Injury
Brief Title: Pediatric Locomotor Training Bladder Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Kosair Charities, Inc. (Other)
Responsible Party: Principal Investigator, Charles Hubscher, Professor, University of Louisville
Other Study IDs: 17.1007
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder
Keywords: Locomotor Training; Urodynamics
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locomotor Training: Assessments for bladder function will be conducted pre-training and following 80 sessions of locomotor training. Locomotor training consists of body-weight supported stepping on a treadmill for one hour.
  Interventions: Procedure: Locomotor Training

INTERVENTIONS:
Procedure: Locomotor Training — Body-weight supported stepping on a treadmill.
  Other Names: Step Training

SUMMARY:
Bladder dysfunction is one of the most important factors influencing duration and quality of life in children with spinal cord injury. Effective bladder control comprises a major aspect of a child's life with SCI and is especially challenging due to the rapid changes in a child's physical and cognitive development. Urological consequences secondary to a neurogenic bladder are responsible for many clinical complications post-spinal cord injury, including repeated urinary tract infections, autonomic dysreflexia, lifelong urologic care, and many hospitalizations. Alternative approaches to bladder management that focus on recovery of function and age-appropriate independence are needed. Prior research findings in our lab in adult participants indicate a benefit of locomotor training on bladder function. The purpose of this study is to determine with quantitative unbiased urodynamic outcome measures if locomotor training, provided to children with spinal cord injury, impacts the developing urinary system.

DETAILED DESCRIPTION:
Our overall hypothesis is that spinal cord injury-induced bladder dysfunction, facilitated by the loss of supra-spinal connections and subsequent alterations of the lumbosacral circuitry, can be ameliorated through activity-based therapy that regulates the state of detrusor-sphincter dyssynergia and normalizes release of neurotrophic factors known to contribute to bladder hyper-reflexia. The primary study aim is to determine the effects of weight-bearing task-specific training for locomotion (stepping on a treadmill) after incomplete and complete spinal cord injury in children on bladder storage, voiding, biomarkers, and quality of life (parent-reported during baseline and exit interview). A secondary aim is to develop a scale for classifying bladder recovery after spinal cord injury based either on the pattern of storage and voiding prior to injury (if the child had bladder control prior to injury) or on established patterns of micturition development (if the child was injured prior to experiencing bladder control).

ELIGIBILITY:
Inclusion Criteria:

* Supra-sacral, non-progressive spinal cord injury
* Bladder dysfunction post-injury

Exclusion Criteria:

* Use of anti-spasticity medications or unwillingness to wean off of medications
* Botox (onabotulinumtoxinA) in the bladder within 9 months of the study
* Bladder dysfunction or urinary tract impairment prior to injury

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children, 2 to 18 years old, who sustained an upper motor neuron spinal cord injury and are medically approved for enrollment in an outpatient, standardized locomotor training program at the University of Louisville (either clinic or research-based) are eligible for participation. Each participant will serve as his/her own control reducing the variability among individuals related to the injury itself, time since injury, medications taken, therapies received, differences in degree of bladder dysfunction, capacity to independently void prior to injury, and many other factors that cannot be controlled in the human experience.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Bladder Storage | 2 years
  Bladder Capacity

SECONDARY OUTCOMES:
Bladder Emptying | 2 years
  Voiding Efficiency
Bladder Pressure | 2 years
  Leak Point and Maximum Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hubscher, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No